CLINICAL TRIAL: NCT01524978
Title: An Open-label, Phase II Study of Vemurafenib in Patients With BRAF V600 Mutation-positive Cancers
Brief Title: A Study of Vemurafenib in Participants With BRAF V600 Mutation-Positive Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MO28072; 2011-004426-10 (EudraCT Number)
Record Dates: First submitted 2012-01-27; First posted 2012-02-02 (Estimated); Results first posted 2017-11-20 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-10

CONDITIONS: Multiple Myeloma, Neoplasms
MeSH Terms: conditions — Multiple Myeloma; Neoplasms | interventions — Cetuximab; Vemurafenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort 1: Non-Small Cell Lung Cancer (NSCLC) - vemurafenib (Experimental): Participants with NSCLC will be treated with vemurafenib monotherapy.
  Interventions: Drug: vemurafenib
- Cohort 2: Ovarian Cancer - vemurafenib (Experimental): Participants with ovarian cancer will be treated with vemurafenib monotherapy.
  Interventions: Drug: vemurafenib
- Cohort 3a: Colorectal Cancer - vemurafenib (Experimental): Participants with colorectal cancer will be treated with vemurafenib monotherapy.
  Interventions: Drug: vemurafenib
- Cohort 3b: Colorectal Cancer - vemurafenib + cetuximab (Experimental): Participants with colorectal cancer will be treated with vemurafenib and cetuximab combination therapy.
  Interventions: Drug: cetuximab; Drug: vemurafenib
- Cohort 4: Cholangiocarcinoma - vemurafenib (Experimental): Participants with cholangiocarcinoma will be treated with vemurafenib monotherapy.
  Interventions: Drug: vemurafenib
- Cohort 6: Multiple Myeloma - vemurafenib (Experimental): Participants with multiple myeloma will be treated with vemurafenib monotherapy.
  Interventions: Drug: vemurafenib
- Cohort 7: Other Solid Tumors - vemurafenib (Experimental): Participants with Erdheim-Chester disease (ECD), Langerhans cell histiocytosis (LCH), anaplastic thyroid cancer, advanced stage astrocytoma, early stage astrocytoma and other BRAF V600-positive tumors will be treated with vemurafenib monotherapy. Subcohorts will be analyzed separately if 7 or more participants are enrolled for each indication.
  Interventions: Drug: vemurafenib

INTERVENTIONS:
Drug: cetuximab — Escalating doses administered on Day 1 and then once weekly by intravenous infusion.
  Arms: Cohort 3b: Colorectal Cancer - vemurafenib + cetuximab
Drug: vemurafenib — Escalating doses given orally twice a day starting on Day 2
  Other Names: Zelboraf
  Arms: Cohort 3b: Colorectal Cancer - vemurafenib + cetuximab
Drug: vemurafenib — 960 mg vemurafenib orally twice a day until disease progression, unacceptable toxicity, or withdrawal of consent.
  Other Names: Zelboraf
  Arms: Cohort 1: Non-Small Cell Lung Cancer (NSCLC) - vemurafenib; Cohort 2: Ovarian Cancer - vemurafenib; Cohort 3a: Colorectal Cancer - vemurafenib; Cohort 4: Cholangiocarcinoma - vemurafenib; Cohort 6: Multiple Myeloma - vemurafenib; Cohort 7: Other Solid Tumors - vemurafenib

SUMMARY:
This open-label, multi-center study will assess the efficacy and safety of vemurafenib in participants with BRAF V600 mutation-positive cancers (solid tumors and multiple myeloma, except melanoma and papillary thyroid cancer) and for whom vemurafenib is deemed the best treatment option in the opinion of the investigator. Participants will receive twice daily oral doses of 960 mg vemurafenib until disease progression, unacceptable toxicity, or withdrawal of consent. The safety and efficacy of vemurafenib in combination with cetuximab in a subset of participants with colorectal cancer will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Must have recovered from all side effects of their most recent systemic or local treatment
* Adequate hematological, renal and liver function

For solid tumors only:

* Histologically confirmed cancers (excluding melanoma and papillary thyroid cancer) with a BRAF V600 mutation and that are resistant to standard therapy or for which standard or curative therapy does not exist
* Measurable disease according to Response Evaluation Criteria In Solid Tumors (RECIST)

For multiple myeloma only:

* Confirmed diagnosis of multiple myeloma with a BRAF V600 mutation
* Must have received at least one prior systemic therapy for the treatment of multiple myeloma
* Treated with local radiotherapy
* Must have relapsed and/or refractory multiple myeloma with measurable disease

Exclusion Criteria:

* Melanoma, papillary thyroid cancer or hematological malignancies (with the exception of multiple myeloma)
* Uncontrolled concurrent malignancy
* Multiple myeloma: solitary bone or solitary extramedullary plasmacytoma as the only evidence of plasma cell dyscrasia
* Active or untreated central nervous system (CNS) metastases
* History of or known carcinomatous meningitis
* Concurrent administration of any anti-cancer therapies other than those administered in this study
* Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that would, in the investigator's opinion, contraindicate participation in this study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2012-04-12 (Actual); Primary Completion 2016-10-28 (Actual); Study Completion 2016-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (34):
- United States (11):
  - Arizona Oncology, Tucson, Arizona
  - Rocky Mountain Cancer Centers, LLP, Aurora, Colorado
  - Massachusetts General Hospital;Oncology, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Vanderbilt, Nashville, Tennessee
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - Yakima Valley Memorial Hospital/North Star Lodge, Yakima, Washington
- Tianjin Cancer Hospital, Tianjin, China
- France (8):
  - Institut Bergonie; Oncologie, Bordeaux
  - Centre Francois Baclesse; Oncologie, Caen
  - Centre Georges François Leclerc, Dijon
  - Centre Leon Berard; Departement Oncologie Medicale, Lyon
  - Institut Paoli-Calmettes; Oncologie Medicale 1, Marseille
  - Centre Rene Gauducheau, Saint-Herblain
  - Institut Claudius Regaud; Departement Oncologie Medicale, Toulouse
  - Institut Gustave Roussy; Sitep, Villejuif
- Germany (3):
  - Klinik der Uni zu Koeln; Klinik I für Innere Medizin; Onkologie, Cologne
  - Universitätsklinikum Essen; Innere Klinik und Poliklinik für Tumorforschung, Essen
  - Universitätsklinikum Mannheim, Tagestherapiezentrum, Interdisziplinäres Tumorzentrum, Mannheim
- Spain (8):
  - Hospital Univ. Central de Asturias; Servicio de Oncologia, Oviedo, Principality of Asturias
  - Hospital del Mar; Servicio de Oncologia, Barcelona
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - Hospital General Universitario Gregorio Marañon; Servicio de Oncologia, Madrid
  - Fundacion Jimenez Diaz; Servicio de Oncologia, Madrid
  - Centro Integral Oncologico Clara Campal (CIOCC); Dirección Médica, Madrid
  - Hospital Clinico Universitario de Salamanca; Servicio de Oncologia, Salamanca
  - Hospital Clinico Universitario de Valencia; Servicio de Onco-hematologia, Valencia
- United Kingdom (3):
  - Aberdeen Royal Infirmary, Aberdeen
  - The Royal Marsden Hospital; Dept of Medicine, London
  - The Royal Marsden Hospital, Sutton

REFERENCES:
- [Derived] Subbiah V, Burris HA 3rd, Kurzrock R. Revolutionizing cancer drug development: Harnessing the potential of basket trials. Cancer. 2024 Jan;130(2):186-200. doi: 10.1002/cncr.35085. Epub 2023 Nov 7. PMID 37934000
- [Derived] Kaley T, Touat M, Subbiah V, Hollebecque A, Rodon J, Lockhart AC, Keedy V, Bielle F, Hofheinz RD, Joly F, Blay JY, Chau I, Puzanov I, Raje NS, Wolf J, DeAngelis LM, Makrutzki M, Riehl T, Pitcher B, Baselga J, Hyman DM. BRAF Inhibition in BRAFV600-Mutant Gliomas: Results From the VE-BASKET Study. J Clin Oncol. 2018 Dec 10;36(35):3477-3484. doi: 10.1200/JCO.2018.78.9990. Epub 2018 Oct 23. PMID 30351999
- [Derived] Hyman DM, Puzanov I, Subbiah V, Faris JE, Chau I, Blay JY, Wolf J, Raje NS, Diamond EL, Hollebecque A, Gervais R, Elez-Fernandez ME, Italiano A, Hofheinz RD, Hidalgo M, Chan E, Schuler M, Lasserre SF, Makrutzki M, Sirzen F, Veronese ML, Tabernero J, Baselga J. Vemurafenib in Multiple Nonmelanoma Cancers with BRAF V600 Mutations. N Engl J Med. 2015 Aug 20;373(8):726-36. doi: 10.1056/NEJMoa1502309. PMID 26287849

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant with breast cancer was screened shortly after Cohort 5 (Breast Cancer) had been closed. This participant was allowed to enter the study in Cohort 7: Other BRAF V600-positive tumors. For analysis purposes Cohort 7 was split into sub-cohorts for indications with sufficient participants.
Groups:
- Cohort 1: Non-Small Cell Lung Cancer (NSCLC) - Vemurafenib: Participants with NSCLC were treated with vemurafenib monotherapy.
- Cohort 2: Ovarian Cancer - Vemurafenib: Participants with ovarian cancer were treated with vemurafenib monotherapy.
- Cohort 3a: Colorectal Cancer - Vemurafenib: Participants with colorectal cancer were treated with vemurafenib monotherapy.
- Cohort 3b: Colorectal Cancer - Vemurafenib + Cetuximab: Participants with colorectal cancer were treated with vemurafenib and cetuximab combination therapy.
- Cohort 4: Cholangiocarcinoma - Vemurafenib: Participants with cholangiocarcinoma were treated with vemurafenib monotherapy.
- Cohort 6: Multiple Myeloma - Vemurafenib: Participants with multiple myeloma were treated with vemurafenib monotherapy.
- Cohort 7a: ECD/LCH - Vemurafenib: Participants with Erdheim-Chester disease (ECD) or Langerhans cell histiocytosis (LCH) were treated with vemurafenib monotherapy.
- Cohort 7b: Anaplastic Thyroid Cancer - Vemurafenib: Participants with anaplastic thyroid cancer were treated with vemurafenib monotherapy.
- Cohort 7c: Advanced Stage Astrocytoma - Vemurafenib: Participants with advanced stage astrocytoma were treated with vemurafenib monotherapy.
- Cohort 7d: Early Stage Astrocytoma - Vemurafenib: Participants with early stage astrocytoma were treated with vemurafenib monotherapy.
- Cohort 7: Other BRAF V600-positive Tumors - Vemurafenib: Participants with other BRAF V600-positive tumors were treated with vemurafenib monotherapy.
Period: Overall Study
Arm/Group | Cohort 1: Non-Small Cell Lung Cancer (NSCLC) - Vemurafenib | Cohort 2: Ovarian Cancer - Vemurafenib | Cohort 3a: Colorectal Cancer - Vemurafenib | Cohort 3b: Colorectal Cancer - Vemurafenib + Cetuximab | Cohort 4: Cholangiocarcinoma - Vemurafenib | Cohort 6: Multiple Myeloma - Vemurafenib | Cohort 7a: ECD/LCH - Vemurafenib | Cohort 7b: Anaplastic Thyroid Cancer - Vemurafenib | Cohort 7c: Advanced Stage Astrocytoma - Vemurafenib | Cohort 7d: Early Stage Astrocytoma - Vemurafenib | Cohort 7: Other BRAF V600-positive Tumors - Vemurafenib
Started | 62 | 4 | 10 | 27 | 9 | 9 | 26 | 12 | 12 | 9 | 28
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 62 | 4 | 10 | 27 | 9 | 9 | 26 | 12 | 12 | 9 | 28
Not completed — Other | 16 | 2 | 1 | 2 | 1 | 3 | 17 | 1 | 2 | 2 | 5
Not completed — Withdrawal by Subject | 12 | 0 | 1 | 1 | 3 | 1 | 6 | 2 | 4 | 0 | 5
Not completed — Lost to Follow-up | 0 | 0 | 3 | 0 | 1 | 1 | 2 | 0 | 1 | 1 | 1
Not completed — Death | 34 | 2 | 5 | 24 | 4 | 4 | 1 | 9 | 5 | 6 | 17

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants enrolled in the study irrespective of whether they had received study medication or not.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Non-Small Cell Lung Cancer (NSCLC) - Vemurafenib | Cohort 2: Ovarian Cancer - Vemurafenib | Cohort 3a: Colorectal Cancer - Vemurafenib | Cohort 3b: Colorectal Cancer - Vemurafenib + Cetuximab | Cohort 4: Cholangiocarcinoma - Vemurafenib | Cohort 6: Multiple Myeloma - Vemurafenib | Cohort 7a: ECD/LCH - Vemurafenib | Cohort 7b: Anaplastic Thyroid Cancer - Vemurafenib | Cohort 7c: Advanced Stage Astrocytoma - Vemurafenib | Cohort 7d: Early Stage Astrocytoma - Vemurafenib | Cohort 7: Other BRAF V600-positive Tumors - Vemurafenib | Total
Number analyzed (Participants) | 62 | 4 | 10 | 27 | 9 | 9 | 26 | 12 | 12 | 9 | 28 | 208
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (10.2) | 45.8 (5.3) | 57.3 (5.4) | 64.3 (8.8) | 53.2 (9.7) | 62.1 (4.3) | 60.8 (13.3) | 66.8 (9.2) | 41.6 (12.2) | 34.3 (20.7) | 53.7 (17.5) | 59.0 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 4 | 5 | 18 | 5 | 3 | 14 | 3 | 8 | 9 | 15 | 111
  Male | 35 | 0 | 5 | 9 | 4 | 6 | 12 | 9 | 4 | 0 | 13 | 97

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Best Overall Response Rate (BORR)
Description: Confirmed BORR: percentage of participants with an objective response (OR) (complete response [CR], partial response [PR], stringent CR [sCR] or very good PR [VGPR]) on 2 occasions >/= 4 weeks apart as assessed by the Investigator using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. or International Myeloma Working Group (IMWG) criteria. RECIST v1.1: CR: disappearance of all target lesions; PR: >/= 30% decrease in the sum of diameters of target lesions. IMWG: CR: negative immunofixation on serum and urine, disappearance of any soft tissue plasmacytomas and </= 5% plasma cells in bone marrow; PR: >/= 50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by >/= 90% or to <200 mg per 24 hours. VGPR: serum and urine M-protein detectable by immunofixation but not on electrophoresis or >/= 90% reduction in serum M-protein plus urine M-protein level < 100 mg per 24 hour; sCR: CR plus normal free light chain (FLC) ratio and no clonal cells in bone marrow.
Time Frame: Up to approximately 3 years
Population: ITT population included all participants enrolled in the study irrespective of whether they had received study drug or not.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Non-Small Cell Lung Cancer (NSCLC) - Vemurafenib | Cohort 2: Ovarian Cancer - Vemurafenib | Cohort 3a: Colorectal Cancer - Vemurafenib | Cohort 3b: Colorectal Cancer - Vemurafenib + Cetuximab | Cohort 4: Cholangiocarcinoma - Vemurafenib | Cohort 6: Multiple Myeloma - Vemurafenib | Cohort 7a: ECD/LCH - Vemurafenib | Cohort 7b: Anaplastic Thyroid Cancer - Vemurafenib | Cohort 7c: Advanced Stage Astrocytoma - Vemurafenib | Cohort 7d: Early Stage Astrocytoma - Vemurafenib | Cohort 7: Other BRAF V600-positive Tumors - Vemurafenib
Number analyzed (Participants) | 62 | 4 | 10 | 27 | 9 | 9 | 26 | 12 | 12 | 9 | 28
percentage of participants | 37.1 [25.16 to 50.31] | 50.0 [6.76 to 93.24] | 0 [0.00 to 30.85] | 7.4 [0.91 to 24.29] | 22.2 [2.81 to 60.01] | 22.2 [2.81 to 60.01] | 61.5 [40.57 to 79.77] | 25.0 [5.49 to 57.19] | 16.7 [2.09 to 48.41] | 33.3 [7.49 to 70.07] | 17.9 [6.06 to 36.89]

2. Secondary Outcome: Percentage of Participants With Confirmed Clinical Benefit
Description: Included were participants with confirmed PR or CR or Stable Disease (SD) that had lasted at least 6 months according to RECIST v1.1 or confirmed CR, PR, VGPR, sCR or SD for at least 6 months according to IMWG criteria. RECIST v1.1: PR: >/= 30% decrease in the sum of diameters of target lesions; CR: disappearance of all target lesions; SD: not meeting criteria for CR, PR or progressive disease (PD). IMWG: CR: negative immunofixation on serum and urine, disappearance of any soft tissue plasmacytomas and </= 5% plasma cells in bone marrow; PR: >/= 50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by >/= 90% or to <200 mg per 24 hours. VGPR: serum and urine M-protein detectable by immunofixation but not on electrophoresis or >/= 90% reduction in serum M-protein plus urine M-protein level < 100 mg per 24 hour; sCR: CR plus normal FLC ratio and no clonal cells in bone marrow; SD: not meeting criteria for CR, VGPR, PR or PD.
Time Frame: Up to approximately 3 years
Population: ITT population included all participants enrolled in the study irrespective of whether they had received study medication or not.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Non-Small Cell Lung Cancer (NSCLC) - Vemurafenib | Cohort 2: Ovarian Cancer - Vemurafenib | Cohort 3a: Colorectal Cancer - Vemurafenib | Cohort 3b: Colorectal Cancer - Vemurafenib + Cetuximab | Cohort 4: Cholangiocarcinoma - Vemurafenib | Cohort 6: Multiple Myeloma - Vemurafenib | Cohort 7a: ECD/LCH - Vemurafenib | Cohort 7b: Anaplastic Thyroid Cancer - Vemurafenib | Cohort 7c: Advanced Stage Astrocytoma - Vemurafenib | Cohort 7d: Early Stage Astrocytoma - Vemurafenib | Cohort 7: Other BRAF V600-positive Tumors - Vemurafenib
Number analyzed (Participants) | 62 | 4 | 10 | 27 | 9 | 9 | 26 | 12 | 12 | 9 | 28
percentage of participants | 48.4 [35.50 to 61.44] | 50.0 [6.76 to 93.24] | 0 [NA to NA] — N/A=NE=not estimable, because of insufficient number of participants with events | 18.5 [6.30 to 38.08] | 44.4 [13.70 to 78.80] | 22.2 [2.81 to 60.01] | 76.9 [56.35 to 91.03] | 25.0 [5.49 to 57.19] | 33.3 [9.92 to 65.11] | 44.4 [13.70 to 78.80] | 17.9 [6.06 to 36.89]

3. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR: percentage of participants with an objective response (OR) (CR, PR, sCR or VGPR) on 2 occasions >/= 4 weeks apart as assessed by the Investigator using RECIST v1.1. or IMWG criteria. RECIST v1.1: CR: disappearance of all target lesions; PR: >/= 30% decrease in the sum of diameters of target lesions. IMWG: CR: negative immunofixation on serum and urine, disappearance of any soft tissue plasmacytomas and </= 5% plasma cells in bone marrow; PR: >/= 50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by >/= 90% or to <200 mg per 24 hours. VGPR: serum and urine M-protein detectable by immunofixation but not on electrophoresis or >/= 90% reduction in serum M-protein plus urine M-protein level < 100 mg per 24 hour; sCR: CR plus normal FLC ratio and no clonal cells in bone marrow.
Time Frame: Up to approximately 3 years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Non-Small Cell Lung Cancer (NSCLC) - Vemurafenib | Cohort 2: Ovarian Cancer - Vemurafenib | Cohort 3a: Colorectal Cancer - Vemurafenib | Cohort 3b: Colorectal Cancer - Vemurafenib + Cetuximab | Cohort 4: Cholangiocarcinoma - Vemurafenib | Cohort 6: Multiple Myeloma - Vemurafenib | Cohort 7a: ECD/LCH - Vemurafenib | Cohort 7b: Anaplastic Thyroid Cancer - Vemurafenib | Cohort 7c: Advanced Stage Astrocytoma - Vemurafenib | Cohort 7d: Early Stage Astrocytoma - Vemurafenib | Cohort 7: Other BRAF V600-positive Tumors - Vemurafenib
Number analyzed (Participants) | 62 | 4 | 10 | 27 | 9 | 9 | 26 | 12 | 12 | 9 | 28
percentage of participants
  CR | 0 [0.00 to 5.78] | 0 [0.00 to 60.24] | 0 [0.00 to 30.85] | 0 [0.00 to 12.77] | 0 [0.00 to 33.63] | 0 [0.00 to 33.63] | 7.7 [0.95 to 25.13] | 8.3 [0.21 to 38.48] | 8.3 [0.21 to 38.48] | 0 [0.00 to 33.63] | 3.6 [0.09 to 18.35]
  PR | 37.1 [25.16 to 50.31] | 50.0 [6.76 to 93.24] | 0 [0.00 to 30.85] | 7.4 [0.91 to 24.29] | 22.2 [2.81 to 60.01] | 11.1 [0.28 to 48.25] | 53.8 [33.37 to 73.41] | 16.7 [2.09 to 48.41] | 8.3 [0.21 to 38.48] | 33.3 [7.49 to 70.07] | 14.3 [4.03 to 32.67]
  VGPR | NA [NA to NA] — N/A= VGPR data only collected in multiple myeloma cohort | NA [NA to NA] — N/A= VGPR data only collected in multiple myeloma cohort | NA [NA to NA] — N/A= VGPR data only collected in multiple myeloma cohort | NA [NA to NA] — N/A= VGPR data only collected in multiple myeloma cohort | NA [NA to NA] — N/A= VGPR data only collected in multiple myeloma cohort | 11.1 [0.28 to 48.25] | NA [NA to NA] — N/A= VGPR data only collected in multiple myeloma cohort | NA [NA to NA] — N/A= VGPR data only collected in multiple myeloma cohort | NA [NA to NA] — N/A= VGPR data only collected in multiple myeloma cohort | NA [NA to NA] — N/A= VGPR data only collected in multiple myeloma cohort | NA [NA to NA] — N/A= VGPR data only collected in multiple myeloma cohort
  sCR | NA [NA to NA] — N/A= sCR data only collected in multiple myeloma cohort | NA [NA to NA] — N/A= sCR data only collected in multiple myeloma cohort | NA [NA to NA] — N/A= sCR data only collected in multiple myeloma cohort | NA [NA to NA] — N/A= sCR data only collected in multiple myeloma cohort | NA [NA to NA] — N/A= sCR data only collected in multiple myeloma cohort | 0 [0.00 to 33.63] | NA [NA to NA] — N/A= sCR data only collected in multiple myeloma cohort | NA [NA to NA] — N/A= sCR data only collected in multiple myeloma cohort | NA [NA to NA] — N/A= sCR data only collected in multiple myeloma cohort | NA [NA to NA] — N/A= sCR data only collected in multiple myeloma cohort | NA [NA to NA] — N/A= sCR data only collected in multiple myeloma cohort

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the period from the date of initial PR or CR for solid tumors according to RECISTv1.1 and CR, PR, VGPR or sCR for multiple myeloma according to IMWG criteria, until the date of PD or death from any cause. RECIST v1.1: PD: At least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. IMWG: PD: increase of >/= 25% from lowest response value in serum or urine M-protein or bone marrow plasma cell percentage or development of new or increase in size of bone lesions or soft tissue plasmacytomas.
Time Frame: Up to approximately 3 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Non-Small Cell Lung Cancer (NSCLC) - Vemurafenib | Cohort 2: Ovarian Cancer - Vemurafenib | Cohort 3a: Colorectal Cancer - Vemurafenib | Cohort 3b: Colorectal Cancer - Vemurafenib + Cetuximab | Cohort 4: Cholangiocarcinoma - Vemurafenib | Cohort 6: Multiple Myeloma - Vemurafenib | Cohort 7a: ECD/LCH - Vemurafenib | Cohort 7b: Anaplastic Thyroid Cancer - Vemurafenib | Cohort 7c: Advanced Stage Astrocytoma - Vemurafenib | Cohort 7d: Early Stage Astrocytoma - Vemurafenib | Cohort 7: Other BRAF V600-positive Tumors - Vemurafenib
Number analyzed (Participants) | 62 | 4 | 10 | 27 | 9 | 9 | 26 | 12 | 12 | 9 | 28
months | 7.16 [5.49 to 18.43] | 8.16 [3.88 to 12.45] | NA [NA to NA] — N/A=NE=not estimable, because of insufficient number of participants with events | 6.54 [5.68 to 7.39] | 12.86 [3.58 to 22.14] | NA [NA to NA] — N/A=NE=not estimable, because of insufficient number of participants with events | NA [NA to NA] — N/A=NE=not estimable, because of insufficient number of participants with events | 9.95 [8.31 to 30.98] | NA [13.08 to NA] — N/A=NE=not estimable, because of insufficient number of participants with events | 3.42 [2.40 to 7.49] | 9.92 [3.48 to 21.22]

5. Secondary Outcome: Time to Response
Description: Time to response was defined as the time from the first day of study treatment to the date of first CR, or PR for solid tumors according to RECISTv1.1 and CR, PR, VGPR or sCR for multiple myeloma according to IMWG criteria. RECIST v1.1: CR: disappearance of all target lesions; PR: at least a 30% decrease in the sum of diameters of target lesions. IMWG criteria: CR: negative immunofixation on serum and urine and disappearance of any soft tissue plasmacytomas and </= 5% plasma cells in bone marrow; PR: >/= 50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by >/= 90% or to < 200 mg per 24 hours. VGPR: serum and urine M-protein detectable by immunofixation but not on electrophoresis or >/= 90% reduction in serum M-protein plus urine M-protein level < 100 mg per 24 hour; sCR: CR plus normal FLC ratio and no clonal cells in bone marrow.
Time Frame: Up to approximately 3 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Non-Small Cell Lung Cancer (NSCLC) - Vemurafenib | Cohort 2: Ovarian Cancer - Vemurafenib | Cohort 3a: Colorectal Cancer - Vemurafenib | Cohort 3b: Colorectal Cancer - Vemurafenib + Cetuximab | Cohort 4: Cholangiocarcinoma - Vemurafenib | Cohort 6: Multiple Myeloma - Vemurafenib | Cohort 7a: ECD/LCH - Vemurafenib | Cohort 7b: Anaplastic Thyroid Cancer - Vemurafenib | Cohort 7c: Advanced Stage Astrocytoma - Vemurafenib | Cohort 7d: Early Stage Astrocytoma - Vemurafenib | Cohort 7: Other BRAF V600-positive Tumors - Vemurafenib
Number analyzed (Participants) | 62 | 4 | 10 | 27 | 9 | 9 | 26 | 12 | 12 | 9 | 28
months | 7.26 [3.68 to NA] — N/A=NE=not estimable due to insufficient number of participants with events | NA [1.64 to NA] — N/A=NE=not estimable due to insufficient number of participants with events | NA [NA to NA] — N/A=NE=not estimable due to insufficient number of participants with events | NA [NA to NA] — N/A=NE=not estimable due to insufficient number of participants with events | NA [3.52 to NA] — N/A=NE=not estimable due to insufficient number of participants with events | 5.75 [NA to NA] — N/A=NE=not estimable due to insufficient number of participants with events | 5.49 [3.68 to 13.73] | NA [1.68 to NA] — N/A=NE=not estimable due to insufficient number of participants with events | NA [1.74 to NA] — N/A=NE=not estimable due to insufficient number of participants with events | NA [2.33 to NA] — N/A=NE=not estimable due to insufficient number of participants with events | NA [3.68 to NA] — N/A=NE=not estimable due to insufficient number of participants with events

6. Secondary Outcome: Time to Tumor Progression (TTP)
Description: TTP was defined as time from the first day of study treatment to the first occurrence of progressive disease (PD). RECIST v1.1: PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. IMWG: PD: increase of >/= 25% from lowest response value in serum or urine M-protein or bone marrow plasma cell percentage or development of new or increase in size of bone lesions or soft tissue plasmacytomas.
Time Frame: Up to approximately 3 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Non-Small Cell Lung Cancer (NSCLC) - Vemurafenib | Cohort 2: Ovarian Cancer - Vemurafenib | Cohort 3a: Colorectal Cancer - Vemurafenib | Cohort 3b: Colorectal Cancer - Vemurafenib + Cetuximab | Cohort 4: Cholangiocarcinoma - Vemurafenib | Cohort 6: Multiple Myeloma - Vemurafenib | Cohort 7a: ECD/LCH - Vemurafenib | Cohort 7b: Anaplastic Thyroid Cancer - Vemurafenib | Cohort 7c: Advanced Stage Astrocytoma - Vemurafenib | Cohort 7d: Early Stage Astrocytoma - Vemurafenib | Cohort 7: Other BRAF V600-positive Tumors - Vemurafenib
Number analyzed (Participants) | 62 | 4 | 10 | 27 | 9 | 9 | 26 | 12 | 12 | 9 | 28
months | 7.33 [5.29 to 9.66] | 6.44 [1.87 to 14.29] | 3.88 [1.84 to 5.52] | 3.68 [3.45 to 5.39] | 3.02 [1.64 to 9.00] | 4.63 [2.89 to NA] — N/A=NE=not estimable due to insufficient number of participants with events | NA [NA to NA] — N/A=NE=not estimable due to insufficient number of participants with events | 2.83 [1.77 to 5.49] | 5.62 [1.81 to 14.85] | 5.36 [3.02 to 9.10] | 3.65 [1.68 to 5.75]

7. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the first day of study treatment, until the first documented PD or death from any cause, whichever occurs first. RECIST v1.1: PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. IMWG criteria: PD: increase of >/= 25% from lowest response value in serum or urine M-protein or bone marrow plasma cell percentage or development of new or increase in size of bone lesions or soft tissue plasmacytomas.
Time Frame: Up to approximately 3 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Non-Small Cell Lung Cancer (NSCLC) - Vemurafenib | Cohort 2: Ovarian Cancer - Vemurafenib | Cohort 3a: Colorectal Cancer - Vemurafenib | Cohort 3b: Colorectal Cancer - Vemurafenib + Cetuximab | Cohort 4: Cholangiocarcinoma - Vemurafenib | Cohort 6: Multiple Myeloma - Vemurafenib | Cohort 7a: ECD/LCH - Vemurafenib | Cohort 7b: Anaplastic Thyroid Cancer - Vemurafenib | Cohort 7c: Advanced Stage Astrocytoma - Vemurafenib | Cohort 7d: Early Stage Astrocytoma - Vemurafenib | Cohort 7: Other BRAF V600-positive Tumors - Vemurafenib
Number analyzed (Participants) | 62 | 4 | 10 | 27 | 9 | 9 | 26 | 12 | 12 | 9 | 28
months | 6.51 [5.16 to 8.97] | 6.44 [1.87 to 14.29] | 3.88 [1.84 to 5.52] | 3.68 [1.81 to 5.39] | 3.02 [1.64 to 9.00] | 4.63 [2.89 to NA] — N/A=NE=not estimable due to insufficient number of participants with events | NA [NA to NA] — N/A=NE=not estimable due to insufficient number of participants with events | 2.83 [1.77 to 5.49] | 9.59 [1.81 to 14.78] | 5.26 [3.02 to 5.72] | 3.12 [1.64 to 5.55]

8. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as time between the first day of study treatment and date of death of any cause.
Time Frame: Up to approximately 3 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Non-Small Cell Lung Cancer (NSCLC) - Vemurafenib | Cohort 2: Ovarian Cancer - Vemurafenib | Cohort 3a: Colorectal Cancer - Vemurafenib | Cohort 3b: Colorectal Cancer - Vemurafenib + Cetuximab | Cohort 4: Cholangiocarcinoma - Vemurafenib | Cohort 6: Multiple Myeloma - Vemurafenib | Cohort 7a: ECD/LCH - Vemurafenib | Cohort 7b: Anaplastic Thyroid Cancer - Vemurafenib | Cohort 7c: Advanced Stage Astrocytoma - Vemurafenib | Cohort 7d: Early Stage Astrocytoma - Vemurafenib | Cohort 7: Other BRAF V600-positive Tumors - Vemurafenib
Number analyzed (Participants) | 62 | 4 | 10 | 27 | 9 | 9 | 26 | 12 | 12 | 9 | 28
months | 15.38 [9.56 to 22.77] | NA [2.56 to NA] — N/A=NE=not estimable due to insufficient number of participants with events | 9.30 [7.82 to 12.88] | 7.16 [5.49 to 11.73] | 17.94 [11.20 to NA] — N/A=NE=not estimable due to insufficient number of participants with events | 24.54 [4.96 to NA] — N/A=NE=not estimable due to insufficient number of participants with events | NA [NA to NA] — N/A=NE=not estimable due to insufficient number of participants with events | 5.88 [2.17 to 16.79] | 40.11 [9.59 to 40.11] | 12.75 [6.70 to NA] — N/A=NE=not estimable due to insufficient number of participants with events | 11.56 [3.71 to 28.16]

9. Secondary Outcome: Maximum Tolerated Dose for Vemurafenib in Combination With Cetuximab
Description: Cohort 3b included participants with colorectal cancer treated with escalating doses of vemurafenib and cetuximab. The escalating doses were as follows: Dose Level 1: 720 milligrams (mg) of vemurafenib orally twice daily starting on Day 2 of Cycle 1 and 300 milligrams per square meter (mg/m^2) loading dose of cetuximab by infusion and then 200 mg/m^2 weekly; Dose Level 2: 720 mg of vemurafenib twice daily starting on Day 2 of Cycle 1 and 400 mg/m^2 loading dose of cetuximab and then 250 mg/m^2 weekly; Dose Level 3: 960 mg of vemurafenib twice daily starting on Day 2 of Cycle 1 and 400 mg/m^2 loading dose of cetuximab and then 250 mg/m^2 weekly. Reported here are the maximum tolerated doses for each vemurafenib and cetuximab.
Time Frame: Up to approximately 3 years
Population: All participants from Cohort 3b who received at least one dose of study medication.
Measure: Number; unit: milligrams (mg)
Arm/Group | Cohort 1: Non-Small Cell Lung Cancer (NSCLC) - Vemurafenib | Cohort 2: Ovarian Cancer - Vemurafenib | Cohort 3a: Colorectal Cancer - Vemurafenib | Cohort 3b: Colorectal Cancer - Vemurafenib + Cetuximab | Cohort 4: Cholangiocarcinoma - Vemurafenib | Cohort 6: Multiple Myeloma - Vemurafenib | Cohort 7a: ECD/LCH - Vemurafenib | Cohort 7b: Anaplastic Thyroid Cancer - Vemurafenib | Cohort 7c: Advanced Stage Astrocytoma - Vemurafenib | Cohort 7d: Early Stage Astrocytoma - Vemurafenib | Cohort 7: Other BRAF V600-positive Tumors - Vemurafenib
Number analyzed (Participants) | 0 | 0 | 0 | 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0
milligrams (mg)
  vemurafenib |  |  |  | 960 |  |  |  |  |  |  |
  cetuximab |  |  |  | 400 |  |  |  |  |  |  |

10. Secondary Outcome: Number of Dose-limiting Toxicities of Vemurafenib in Combination With Cetuximab
Description: Cohort 3b included participants with colorectal cancer treated with escalating doses of vemurafenib and cetuximab. The escalating doses were as follows: Dose Level 1: 720 milligrams (mg) of vemurafenib orally twice daily starting on Day 2 of Cycle 1 and 300 milligrams per square meter (mg/m^2) loading dose of cetuximab by infusion and then 200 mg/m^2 weekly; Dose Level 2: 720 mg of vemurafenib twice daily starting on Day 2 of Cycle 1 and 400 mg/m^2 loading dose of cetuximab and then 250 mg/m^2 weekly; Dose Level 3: 960 mg of vemurafenib twice daily starting on Day 2 of Cycle 1 and 400 mg/m^2 loading dose of cetuximab and then 250 mg/m^2 weekly. Reported here are type and number of dose limited toxicities observed.
Time Frame: Up to 28 days
Population: All participants from Cohort 3b who received at least one dose of study medication.
Measure: Number; unit: dose-limiting toxicities
Arm/Group | Cohort 1: Non-Small Cell Lung Cancer (NSCLC) - Vemurafenib | Cohort 2: Ovarian Cancer - Vemurafenib | Cohort 3a: Colorectal Cancer - Vemurafenib | Cohort 3b: Colorectal Cancer - Vemurafenib + Cetuximab | Cohort 4: Cholangiocarcinoma - Vemurafenib | Cohort 6: Multiple Myeloma - Vemurafenib | Cohort 7a: ECD/LCH - Vemurafenib | Cohort 7b: Anaplastic Thyroid Cancer - Vemurafenib | Cohort 7c: Advanced Stage Astrocytoma - Vemurafenib | Cohort 7d: Early Stage Astrocytoma - Vemurafenib | Cohort 7: Other BRAF V600-positive Tumors - Vemurafenib
Number analyzed (Participants) | 0 | 0 | 0 | 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0
dose-limiting toxicities
  Grade 3 amylase increased |  |  |  | 1 |  |  |  |  |  |  |
  Grade 4 lipase increased |  |  |  | 1 |  |  |  |  |  |  |

11. Secondary Outcome: Safety: Percentage of Participants With Adverse Event
Description: An adverse event is any untoward medical occurrence in a subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Up to approximately 3 years
Population: The safety population included all participants who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Non-Small Cell Lung Cancer (NSCLC) - Vemurafenib | Cohort 2: Ovarian Cancer - Vemurafenib | Cohort 3a: Colorectal Cancer - Vemurafenib | Cohort 3b: Colorectal Cancer - Vemurafenib + Cetuximab | Cohort 4: Cholangiocarcinoma - Vemurafenib | Cohort 6: Multiple Myeloma - Vemurafenib | Cohort 7a: ECD/LCH - Vemurafenib | Cohort 7b: Anaplastic Thyroid Cancer - Vemurafenib | Cohort 7c: Advanced Stage Astrocytoma - Vemurafenib | Cohort 7d: Early Stage Astrocytoma - Vemurafenib | Cohort 7: Other BRAF V600-positive Tumors - Vemurafenib
Number analyzed (Participants) | 62 | 4 | 10 | 27 | 9 | 9 | 26 | 12 | 12 | 9 | 28
percentage of participants | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 91.7 | 100 | 100 | 100

ADVERSE EVENTS:
Time Frame: From baseline up to approximately 3 years
Description: The safety population included all participants who received at least one dose of study medication.
Groups:
- Pooled Arm - Vemurafenib: Participants with a variety of cancer types, who were treated with vemurafenib monotherapy, were combined into this arm.
Arm/Group | Cohort 3b: Colorectal Cancer - Vemurafenib + Cetuximab | Pooled Arm - Vemurafenib
Serious Adverse Events (participants affected / at risk) | 11/27 | 91/181
Other Adverse Events (participants affected / at risk) | 26/27 | 177/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 3b: Colorectal Cancer - Vemurafenib + Cetuximab (N=27) | Pooled Arm - Vemurafenib (N=181)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 25
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 18
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 7
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Subileus (Gastrointestinal disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 2
Cholestasis (Hepatobiliary disorders) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 4
Bladder dilatation (Renal and urinary disorders) | 1 | 0
Obstructive uropathy (Renal and urinary disorders) | 1 | 0
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Paraganglion neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Sepsis (Infections and infestations) | 0 | 6
Pneumonia (Infections and infestations) | 0 | 5
Lung infection (Infections and infestations) | 0 | 4
Bronchitis (Infections and infestations) | 0 | 3
Lower respiratory tract infection (Infections and infestations) | 0 | 2
Abdominal abscess (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Furuncle (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Laryngeal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Partial seizures (Nervous system disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Fatigue (General disorders) | 0 | 2
Chest pain (General disorders) | 0 | 1
Hyperthermia (General disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 3
Acute coronary syndrome (Cardiac disorders) | 0 | 2
Pericarditis (Cardiac disorders) | 0 | 2
Dressler's syndrome (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Duodenal perforation (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Pseudolymphoma (Blood and lymphatic system disorders) | 0 | 1
Splenic infarction (Blood and lymphatic system disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Iridocyclitis (Eye disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Body temperature increased (Investigations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 3b: Colorectal Cancer - Vemurafenib + Cetuximab (N=27) | Pooled Arm - Vemurafenib (N=181)
Anaemia (Blood and lymphatic system disorders) | 3 | 30
Abdominal pain (Gastrointestinal disorders) | 12 | 12
Abdominal pain upper (Gastrointestinal disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 5 | 26
Diarrhoea (Gastrointestinal disorders) | 13 | 49
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Flatulence (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 9 | 54
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0
Stomatitis (Gastrointestinal disorders) | 4 | 19
Vomiting (Gastrointestinal disorders) | 8 | 41
Asthenia (General disorders) | 10 | 39
Chest pain (General disorders) | 2 | 0
Chills (General disorders) | 2 | 10
Fatigue (General disorders) | 6 | 60
Oedema peripheral (General disorders) | 4 | 21
Pyrexia (General disorders) | 5 | 26
Conjunctivitis (Infections and infestations) | 3 | 0
Folliculitis (Infections and infestations) | 3 | 18
Oral candidiasis (Infections and infestations) | 2 | 0
Rash pustular (Infections and infestations) | 3 | 0
Skin infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 3 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0
Sunburn (Injury, poisoning and procedural complications) | 4 | 22
Amylase increased (Investigations) | 6 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 15
Blood bilirubin increased (Investigations) | 3 | 10
Electrocardiogram QT prolonged (Investigations) | 4 | 37
Lipase increased (Investigations) | 9 | 10
Lymphocyte count decreased (Investigations) | 3 | 0
Weight decreased (Investigations) | 6 | 20
Decreased appetite (Metabolism and nutrition disorders) | 10 | 50
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 18
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 79
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 18
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 18
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 13
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 41
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 36
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 50
Headache (Nervous system disorders) | 4 | 26
Anxiety (Psychiatric disorders) | 2 | 14
Depression (Psychiatric disorders) | 3 | 10
Haematuria (Renal and urinary disorders) | 2 | 0
Micturition urgency (Renal and urinary disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 31
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 22
Actinic keratosis (Skin and subcutaneous tissue disorders) | 4 | 28
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 57
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 39
Erythema (Skin and subcutaneous tissue disorders) | 7 | 24
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 4 | 58
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 5 | 39
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 42
Rash (Skin and subcutaneous tissue disorders) | 10 | 44
Rash generalised (Skin and subcutaneous tissue disorders) | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 42
Skin fissures (Skin and subcutaneous tissue disorders) | 2 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 2 | 0
Hypertension (Vascular disorders) | 3 | 28
Dry eye (Eye disorders) | 0 | 11
Dry mouth (Gastrointestinal disorders) | 0 | 12
Dysphagia (Gastrointestinal disorders) | 0 | 14
Cyst (General disorders) | 0 | 21
Xerosis (General disorders) | 0 | 16
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 11
Alanine aminotransferase increased (Investigations) | 0 | 15
Blood alkaline phosphatase increased (Investigations) | 0 | 11
Blood creatinine increased (Investigations) | 0 | 19
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 14
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 17
Dysgeusia (Nervous system disorders) | 0 | 24
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 27
Insomnia (Psychiatric disorders) | 0 | 18
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 10
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 18
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 10
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 0 | 33
Milia (Skin and subcutaneous tissue disorders) | 0 | 16
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 48
Papule (Skin and subcutaneous tissue disorders) | 0 | 13
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 21
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.